CLINICAL TRIAL: NCT03649620
Title: A 12-week, Randomized, Double-blind, Placebo-controlled Human Trial to Evaluate the Efficacy and Safety of Unripe Bokbunja Extract on Improvement of Blood Cholesterol
Brief Title: Efficacy and Safety of Unripe Bokbunja Extract on Improvement of Blood Cholesterol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Jong Ho Lee, Professor, Principal Investigator, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BC_cholesterol
Record Dates: First submitted 2018-07-30; First posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-05

CONDITIONS: Blood Cholesterol
Keywords: cholesterol; Bokbunja; Clinical Trial

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- unripe Bokbunja Extract (Experimental): tablet(1 tablet/d, 600 mg/d) for 12 weeks
  Interventions: Dietary Supplement: unripe Bokbunja Extract; Dietary Supplement: Placebo
- Placebo (Placebo Comparator): Placebo for 12 weeks
  Interventions: Dietary Supplement: unripe Bokbunja Extract; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: unripe Bokbunja Extract — tablet(1 tablet/d, 600 mg/d) for 12 weeks
Dietary Supplement: Placebo — Placebo for 12 weeks

SUMMARY:
This study was conducted to investigate the effects of daily supplementation of unripe Bokbunja extract on improvement of blood cholesterol.

DETAILED DESCRIPTION:
This study was a 12 weeks, randomized, double-blind, placebo-controlled human trial. Forty subjects were randomly divided into unripe Bokbunja extract 600 mg or placebo group. The investigators measured total cholesterol, lipid profile, arteriosclerosis index, anthropometric index, oxidized LDL.

ELIGIBILITY:
Inclusion Criteria:

* age between 20 and 65 years,
* Total cholesterol 200-239 mg/dl
* subjects giving written informed consent

Exclusion Criteria:

* Cardiovascular disease, e.g. arrhythmia, heart failure, myocardial infarction
* History of disease that could interfere with the test products or impede their absorption, such as gastrointestinal disease or gastrointestinal surgery
* Participation in any other clinical trials within past 2 months
* Laboratory test, medical or psychological conditions deemed by the investigators to interfere with successful participation in the study
* Pregnancy or breast feeding etc,.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Changes of Total cholesterol | 12 weeks
  Changes of total cholesterol were assessed before and after the intervention

SECONDARY OUTCOMES:
Changes of Lipid profile(total cholesterol, LDL-cholesterol, triglyceride, HDL-cholesterol, free fatty acid, Apolipoprotein A1, Apolipoprotein B, Lipoprotein a, hs-CRP) | 12 weeks
  Changes of lipid profile(total cholesterol, LDL-cholesterol, triglyceride, HDL-cholesterol, free fatty acid, Apolipoprotein A1, Apolipoprotein B, Lipoprotein a, hs-CRP) were assessed before and after the intervention
Changes of Arteriosclerosis index(total cholesterol/HDL-cholesterol, LDL-cholesterol/HDL-cholesterol, triglyceride/HDL-cholesterol, (total HDL-cholesterol-HDL-cholesterol)/HDL-cholesterol, Apolipoprotein B/Apolipoprotein A1) | 12 weeks
  Changes of arteriosclerosis index(total cholesterol/HDL-cholesterol, LDL-cholesterol/HDL-cholesterol, triglyceride/HDL-cholesterol, (total HDL-cholesterol-HDL-cholesterol)/HDL-cholesterol, Apolipoprotein B/Apolipoprotein A1) were assessed before and after the intervention
Changes of Anthropometric index(weight, body mass index, waist hip ratio, waist, hip, fat percentage, lean body mass) | 12 weeks
  Changes of anthropometric index(weight, body mass index, waist hip ratio, waist, hip, fat percentage, lean body mass) were assessed before and after the intervention
Changes of Oxidized LDL | 12 weeks
  Changes of oxidized LDL were assessed before and after the intervention

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cho JM, Chae J, Jeong SR, Moon MJ, Ha KC, Kim S, Lee JH. The cholesterol-lowering effect of unripe Rubus coreanus is associated with decreased oxidized LDL and apolipoprotein B levels in subjects with borderline-high cholesterol levels: a randomized controlled trial. Lipids Health Dis. 2020 Jul 9;19(1):166. doi: 10.1186/s12944-020-01338-z. PMID 32646501